CLINICAL TRIAL: NCT03642613
Title: A Non-interventional, Cross-sectional Study for Evaluating Factors Relating to Daily Step Counts and Physical Activity in Japanese Patients With COPD.
Brief Title: The Study for Evaluating Factors Relating to Daily Step Counts and Physical Activity in Japanese Patients With COPD.
Acronym: STEP-COPD
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Collaborators: Linical Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: D5980R00006
Record Dates: First submitted 2018-08-09; First posted 2018-08-22 (Actual); Last update posted 2020-09-14 (Actual); Status verified 2020-09

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: COPD, RWE, Physical Activity
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Weeks
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is conducted as a multicenter, non-interventional, cross-sectional study. Patients will be enrolled in the study by a continuous registration method after patients provide written informed consent. After providing informed consent, patients will answer the questionnaires and start measurement with an accelerometer within four weeks. Activities will be measured for 14 consecutive days.

DETAILED DESCRIPTION:
This study is conducted as a multicenter, non-interventional, cross-sectional study. Patients will be enrolled in the study by a continuous registration method after patients provide written informed consent. After providing informed consent, patients will answer the questionnaires and start measurement with an accelerometer within four weeks. Activities will be measured for 14 consecutive days.

<Objectives>

* Evaluation of factors relating to physical activity level in COPD patients.
* Evaluation of the number of daily steps in subgroups of COPD patients grouped according to patient characteristics including lung functions, mMRC, and CAT scores.
* Elucidation of impacts of factors associating PAL in COPD patients.
* Elucidating exploratorily the characteristics of the patients who are distributed differently in each factor and analyzing patients' PAL further with their background.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who have provided written informed consent for participation in this study
2. Male and female patients aged at least 40 years at the time of enrolment who are given diagnosis of COPD by a physician*1
3. Patients whose respiratory function test values after bronchodilators (FEV1, FVC, IC) are available*2
4. Patients whose DLCO values and data on the presence/absence of emphysema by a chest CT scan are available*3
5. Outpatients who are able to answer the questionnaires and start measurement with an activity meter within four weeks after informed consent and measure activities for 14 consecutive days

   * 1: Guideline 12) should be referenced for the diagnostic criteria of COPD.
   * 2: Patients whose respiratory function test values after bronchodilators at the time of enrolment or within three months prior to enrolment are available. For patients on a bronchodilator as a long-term controller, respiratory function test values after bronchodilator in the morning of the test are acceptable.
   * 3: This refers to patients who have undergone tests within past one year.

Exclusion Criteria:

1. Patients who have participated in any other interventional studies such as clinical trials within the past eight weeks
2. Patients determined to be inappropriate to be enrolled in this study by investigators because they cannot comply with the procedures, limitations, and requirements of this study, or for other reasons.
3. Patients with an exacerbation of COPDa within the past eight weeks a Exacerbation of COPD: Conditions with increased shortness of breath, increased cough and sputum, occurrence of chest discomfort/uneasiness or its intensification, and which require changes in treatment on disease stable state, excluding cases where there is any other precedent disease (heart failure, pneumothorax, pulmonary thromboembolism, etc.).
4. Patients who require home oxygen therapy (excluding those who use it only during nighttime)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 1. Patients who have provided written informed consent for participation in this study
  2. Male and female patients aged at least 40 years at the time of enrolment who are given diagnosis of COPD by a physician (forced expiratory volume in one second/forced vital capacity [FEV1/FVC] of <70% after bronchodilators within the past one year or at the time of enrolment)
  3. Patients whose respiratory function test values after bronchodilators are available
  4. Patients whose DLCO values and data on the presence/absence of emphysema by a chest CT scan are available
  5. Outpatients who are able to answer the questionnaires and start measurement with an activity meter within four weeks after informed consent and measure activities for 14 consecutive days
Sampling Method: Non-Probability Sample
Enrollment: 505 (Actual)
Dates: Start 2018-09-14 (Actual); Primary Completion 2019-03-15 (Actual); Study Completion 2019-03-15 (Actual)

PRIMARY OUTCOMES:
Physical activity level | 2 weeks
  Physical activity level will be assessed as average daily duration (min) of ≧2 metabolic equivalents (METs)

CONTACTS AND LOCATIONS:
Overall Officials: Masakazu Ichinose, Professor, Study Chair — Tohoku University School of Medicine
Locations (1):
- Tohoku University School of Medicine, Sendai, Miyagi, Japan

REFERENCES:
- [Derived] Ichinose M, Minakata Y, Motegi T, Takahashi T, Seki M, Sugaya S, Hayashi N, Kuwahira I. A Non-Interventional, Cross-Sectional Study to Evaluate Factors Relating to Daily Step Counts and Physical Activity in Japanese Patients with Chronic Obstructive Pulmonary Disease: STEP COPD. Int J Chron Obstruct Pulmon Dis. 2020 Dec 22;15:3385-3396. doi: 10.2147/COPD.S277782. eCollection 2020. PMID 33376319
- See also: CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5980R00006&attachmentIdentifier=a7df13ff-53ca-4862-bd37-880c9b4f308c&fileName=STEP_CSR_Synopsis_Fix.pdf&versionIdentifier=